CLINICAL TRIAL: NCT01369797
Title: Prospective Randomized Study of the Impact on the Autonomy of the Elderly of 75 Years of Age and Older by the Unit for Prevention, Monitoring and Analysis of Aging (UPSAV).
Brief Title: Prospective Randomized Study of the Impact on the Autonomy of the Elderly of 75 Years of Age and Older by the UPSAV
Acronym: GEROPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I10010
Record Dates: First submitted 2011-05-16; First posted 2011-06-09 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: the Elderly of 75 Years and Older Living at Home
Keywords: UPSAV; autonomy; the elderly of 75 years and older

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- reference (No Intervention): "reference" group, where every patient will benefit: of the same GGA at home as those of the " specific intervention " group. The GGA results will not be supplied to the family practioner.
- specific intervention (Experimental): "specific intervention" group, where every patient will benefit: of an GGA at home. According to the frailties or the detected morbidity, a specific plan of intervention will be established for the person. all the preventive actions will be coordinated by UPSAV.
  Interventions: Other: specific intervention

INTERVENTIONS:
Other: specific intervention — Patients included in the "specific intervention" group will benefit from a personalized action plan presented in a multidisciplinary staff that will be established according to the detected frailties. In follow up visits, a new evaluation will be done and the action plan reviewed.
  Arms: specific intervention

SUMMARY:
Background :

The evolving concept of frailty was born in the United States under the term of " frail elderly ". It allows describing geriatrics situations, dominated by the weakness or the functional instability of aged person, illustrating situations at risk. It is about an effective concept, especially in the field of the prevention where it determines strategies of specific care. The ageing, changing according to individuals, is characterized by a decrease of the physiological reserves leading to a precarious balance and to a destabilization.

Epidemiological studies show a very uneven distribution of three categories of old persons according to their health status. Every year, approximately, 12 % of the independent population of 75 years of age and older and living at home, lose their autonomy for one of the activities of the daily life and turn into frailty.

Identifying frailty of old subjects is interesting in order to apply preventive and specific care strategies to reduce the risks of decompensation. The Global Geriatric Assessment (GGA) is the gold standard to detect frailty in this population. The beneficial effects of the GGA during the hospitalization have been recognized in international literature.

The ageing heterogeneousness complexity and the high time-consuming character of GGA led to a difficult approach for the nurses or family practioners in taking care of old persons at home.

To balance these difficulties and to optimize prevention of dependence in the elderly, an experimental unit of prevention was created : Unit for Prevention, Monitoring and Analysis of Aging (UPSAV) on January 4th, 2010 within the geriatric department of the Hospital University of Limoges. It is an innovative organizational structure because, for the first time, the geriatric expertise is proposed freely to the elderly at home. A multidisciplinary gerontological team consisting in a geriatrician, a nurse, a psychomotor therapist and an occupational therapist, can, on requiry, move at old persons' home to make a preventive GGA to detect the risks of loss of autonomy and to propose a coordination of preventive actions.

Purpose :

UPSAV's endpoints are to prevent frail elderly persons from the risk of autonomy loss. This action is led in partnership with all the professionals working around old persons.

The randomized study endpoint is to evaluate elderly from 75 years of age and older at home and to select two homogeneous groups: "reference" and " specific intervention ".

DETAILED DESCRIPTION:
Abstract : The recruitment will be made in the Limousin region within a period of one year by cooptation of families, patients, family practitioners and other partners.

After checking the inclusion criteria and obtaining the signatures of consents, patients will be assessed using the functional status (SMAF) and the Global Geriatric Assessment (GGA).

Patients included in the "specific intervention" group will benefit from a personalized action plan presented in a multidisciplinary staff that will be established according to the detected frailties. In follow up visits, a new evaluation will be done and the action plan reviewed.

Every month, patients of this group will receive a Unit for Prevention, Monitoring and Analysis of Aging (UPSAV) phone call in order to complete the secondary assessment criteria of the trial. Therefore, every patient will be re-evaluated according to the intervention plan of the study.

The quality of life of the patient will be estimated by the scale EQ-5D. In every visit, will be collected in a forward-looking way the medical direct costs (ambulatory, hospital care and medicines) and the non medical costs (transport, helpers, arrangements of the place of residence).

ELIGIBILITY:
Inclusion Criteria:

* 75 years of age and older man or woman
* Patient covered by the health care system
* Patient coverd by a complementary health system or supported by 100% by the health care system
* Patient having the intellectual skills to understand the study, to respect its imperatives and accept the UPSAV's plan or subject with mild to moderate dementia (MMSE > 10) but with a caregiver at home capable of understanding the protocol and of making respect its imperatives written consent signed by the patient

Exclusion Criteria:

* Nursing-home resident
* Mild to moderate dementia (MMSE > 10) without caregiver
* Severe dementia (MMSE < 10)
* Diseases with vital short-term endpoint

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 440 (Actual)
Dates: Start 2011-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Increase of 5 points of the score(function status) SMAF in 2 years | 2 years
  To evaluate at 2 years the impact of the preventive and coordination action of the UPSAV's gerontological expertise by means of a questionnaire of quality of life.

SECONDARY OUTCOMES:
Evaluation of the mortality in 2 years | 2 years
  At 2 years:
  To evaluate the impact on the mortality of the intervention of UPSAV on the studied population.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DANTOINE, Principal Investigator — Limoges UH
Locations (1):
- Pôle Personnes âgées et soins à domicile - Limoges UH, Limoges, Limoges, France